CLINICAL TRIAL: NCT06031727
Title: A Trial to Evaluate the Safety, Tolerability, and Efficacy of CRISPR-Cas13 RNA-editing Therapy Targeting Knockdown of Vascular Endothelial Growth Factor a (HG202) in the Treatment of Neovascular Age-related Macular Degeneration (nAMD)
Brief Title: CRISPR/cas13-medIated RNA TarGeting THerapy for the Treatment of Neovascular Age-related Macular Degeneration Investigator-initiated Trial (SIGHT-I)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: HuidaGene Therapeutics Co., Ltd. (Industry)
Collaborators: Tianjin Medical University Eye Hospital (Other); Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HG20201
Record Dates: First submitted 2023-09-01; First posted 2023-09-11 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Neovascular Age-related Macular Degeneration(nAMD)
Keywords: Macular Degeneration/nAMD/wAMD/Gene-editing/CRISPR/HG202

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HG202 (Experimental)
  Interventions: Genetic: HG202

INTERVENTIONS:
Genetic: HG202 — Method of Administration: Once unilateral subretinal injection; The duration of the study is about 52 weeks for each subject including a 4 weeks screening period, enrollment/baseline visit, treatment visit and 48 weeks follow-up period.

SUMMARY:
Age-related macular degeneration (AMD) is a progressive disease leading to severe and irreversible vision loss of which the neovascular AMD (nAMD) accounted for 90% blindness in AMD. nAMD is primarily driven by the perturbation of vascular endothelial growth factor (VEGF). VEGF overexpression leads to abnormal growth of choroidal neovascularization (CNV), which is a hallmark of AMD. Although anti-VEGF agents are effective in treating nAMD, long-term efficacy decreases over time due to the need for repeated injections impacting patient compliance with treatment regimen while patients still may lose vision during the 7th or 8th year of treatment. These frequent intravitreal injections can increase the risk of complications, including submacular hemorrhage, intraocular hypertension, inflammation, and retinal detachment. Furthermore, there are up to 46% of nAMD patients using anti-VEGF agents who have shown poor response or have developed tachyphylaxis with anti-VEGF therapies. HG202 is a CRISPR/Cas13 RNA-editing therapy packaging novel high-fidelity Cas13 technology using one single AAV vector to partially knock-down the expression of VEGFA and thus inhibit CNV formation in AMD patients who are either responsive or non-responsive to anti-VEGF agents. The long-term, stable delivery of HG202 following a one (1) time gene-editing therapy treatment for nAMD could potentially reduce the frequent injection treatment burden of currently available therapies AND treat nAMD patients who are non-responsive to anti-VEGF therapies and have no treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥ 50 and ≤ 80 years at the time of signing the ICF
* Diagnosed of choroidal neovascularization (CNV) secondary to AMD in the study eye;
* Best-corrected visual acuity (BCVA) ranged from 73 to 23 early treatment diabetic retinopathy study (ETDRS)letter score (corresponding to 20/32 to 20/320 of Snellen visual acuity) in the study eye;
* BCVA in the non-study eye had an ETDRS letter score of 19(equivalent to Snellen visual acuity20/400) and above;
* Able to perform visual acuity and retinal function tests and able and willing to comply with study procedures for this clinical trial;

RESPONSIVE SUBJECTS:

* History of need for and responsive to anti-VEGF therapy in the study eye

NON-RESPONSIVE SUBJECTS:

* History of receiving anti-VEGF therapy but is resistant to treatment, which is defined as: a. complete or near-complete remission of subretinal fluid after the initial 3 doses of anti-VEGF agents and thenno improvement (less than 50um reduction) or deterioration of CRT by OCT

Exclusion Criteria:

* Subretinal hemorrhage, scarring, or fibrosis of greater than 50% of the total lesion in the study eye;
* Any condition in the Investigator's opinion that could limit visual improvement in the study eye;
* Other ocular diseases that may affect central vision in the study eye (e.g., retinal vein occlusion, retinal detachment, macular hole, optic nerve disease, etc.);
* Presence of CNV not due to nAMD in the study eye,
* Uncontrolled glaucoma in the study eye;
* Active intraocular inflammation or a history of uveitis in either eye;
* History or presence of corneal dystrophy in the study eye;
* Subjects with immunodeficiency diseases prone to opportunistic infections;
* History of other intraocular surgery in the study eye within 3 months prior to baseline that in the Investigator's opinion could impact healing or study outcome interpretation;
* Prior gene therapy or oligonucleotide therapy;
* History of acute coronary syndrome, myocardial infarction, coronary revascularization, cerebrovascular accident, or transient ischemic attack within 6 months prior to the Screening Visit;
* Other conditions judged by the investigator as inappropriate for the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of ocular and systemic adverse events | 24 weeks
  Number of adverse events (AEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Incidence and severity of ocular and systemic adverse events | 48 weeks
  Number of adverse events (AEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs)
Change from baseline in best-corrected visual acuity (BCVA) | 24 and 48 weeks
  Change from baseline in BCVA as measured by Early Treatment Diabetic Retinopathy Study (ETDRS) chart in the study eye at different doses
Change from baseline in central retinal thickness (CRT) | 24 and 48 weeks
  Change from baseline in central retinal thickness (CRT) as measured by optical coherence tomography (OCT) in the study eye at different doses
Change From baseline in annualized rate of supplemental injections | 48 weeks
  Change from baseline in the number of anti-VEGF injections which is annualized to a per year rate in the study eye at different doses

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Huidagene Therapeuticd Co., Ltd.
Locations (2):
- China (2):
  - Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical University Eye Hospital, Tianjin, Tianjing

IPD SHARING:
Plan to Share IPD: No